CLINICAL TRIAL: NCT07329764
Title: Effectiveness of a Virtual Reality Intervention on Pain, Anxiety, and Satisfaction in Laboring Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wan-Lin Pan (Other)
Collaborators: Saint Paul's Hospital, Congregation Of The Sisters Of Saint Paul De Chartres (Other)
Responsible Party: Sponsor-Investigator, Wan-Lin Pan, professor, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TYGH114028
Record Dates: First submitted 2025-12-16; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Relieve Pain; Anxiety; Childbirth Experience
Keywords: Virtual Reality; Labor Pain; Anxiety; Childbirth Satisfaction; Non-pharmacological Pain Management; Intrapartum Care
MeSH Terms: conditions — Anxiety Disorders; Labor Pain | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, parallel-group interventional design. Eligible laboring women will be randomly assigned to either a virtual reality (VR) intervention group or a control group with no intervention.
  Participants in the VR group will receive virtual reality-based supportive care during labor, while participants in the control group will receive standard intrapartum care without additional intervention.
  Outcomes will be assessed and compared between the two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Virtual Reality Intervention (Experimental): Participants assigned to this group will receive a virtual reality (VR) intervention during labor.
  The VR intervention consists of immersive natural imagery and music delivered through a head-mounted display as supportive care during labor.
  Interventions: Diagnostic Test: Virtual Reality
- Control: Standard Intrapartum Care (No Intervention): Participants assigned to this group will receive standard intrapartum care without any additional virtual reality intervention.

INTERVENTIONS:
Diagnostic Test: Virtual Reality — Virtual reality interventions offer a promising avenue for addressing the challenges faced by laboring women in Taiwan, particularly in the context of nursing shortages. By effectively reducing pain, anxiety, and improving childbirth satisfaction, these interventions present a cost-effective and easily implementable solution with multiple benefits.
  Arms: Experimental: Virtual Reality Intervention

SUMMARY:
This study is designed to evaluate whether a virtual reality (VR) intervention can help reduce pain and anxiety and improve childbirth satisfaction among laboring women.

Eligible participants will be randomly assigned to either a VR intervention group or a control group receiving standard intrapartum care. Women in the VR group will use a virtual reality headset that provides immersive natural imagery and music during labor, while women in the control group will receive routine care without VR.

The study will compare levels of labor pain, anxiety, and childbirth satisfaction between the two groups to determine the effectiveness of the virtual reality intervention as supportive care during labor.

DETAILED DESCRIPTION:
This randomized, parallel-group interventional study aims to evaluate the effectiveness of a virtual reality (VR) intervention as supportive care during labor. The study will be conducted among laboring women admitted for childbirth who meet the eligibility criteria.

Eligible participants will be randomly assigned to one of two groups: a virtual reality intervention group or a control group receiving standard intrapartum care without additional intervention. Randomization will be performed using an appropriate allocation method to ensure comparable groups. Due to the nature of the intervention, this study will be conducted as an open-label trial.

Participants assigned to the VR intervention group will receive virtual reality-based supportive care during labor. The intervention involves the use of a head-mounted VR device providing immersive natural imagery and calming music, intended to promote relaxation and distraction from labor-related discomfort. The VR intervention will be administered during the active phase of labor according to the study protocol.

Participants in the control group will receive routine intrapartum care in accordance with standard clinical practice, without exposure to virtual reality or other additional supportive interventions beyond usual care.

The primary outcome of the study is labor pain intensity, assessed using the Visual Analogue Scale (VAS) during the active phase of labor. Secondary outcomes include maternal anxiety during labor, measured using the State subscale of the State-Trait Anxiety Inventory (STAI-S), and childbirth satisfaction, assessed using the Childbirth Experience Questionnaire (CEQ) within 48 hours postpartum.

Outcome measures will be compared between the intervention and control groups to determine the effectiveness of the virtual reality intervention in reducing labor pain and anxiety and improving childbirth satisfaction.

ELIGIBILITY:
Women meeting the following criteria were eligible for enrollment:

1. Pregnant.
2. Aged 18 years or older.
3. Pregnant for more than 37 weeks.
4. Single baby born in the cephalic presentation and willing to deliver naturally.
5. Admitted to the hospital during the latent period.
6. No major medical conditions or complications during pregnancy for either mother or baby.
7. Able to hear, speak, read, and write Chinese.
8. Interested in participating in this study and agreeing to complete the questionnaire.

Women meeting the above criteria will be enrolled after the researchers explain the research methods and objectives. Exclusion criteria include:

1. Virtual reality sickness.
2. Vision or hearing problems.
3. Withdrawal from the study.
4. Maternal or fetal condition requiring emergency cesarean section.
5. Those diagnosed with migraine, epilepsy, or mental illness.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Labor pain intensity as measured by the Visual Analogue Scale (VAS) | During the active phase of labor
  Labor pain intensity will be assessed using the Visual Analogue Scale (VAS), a 10-cm horizontal line ranging from 0 (no pain) to 10 (worst imaginable pain).
  Pain scores will be recorded at predefined time points during the active phase of labor.
  Mean VAS scores will be calculated and compared between groups.

SECONDARY OUTCOMES:
Maternal anxiety during labor as measured by the State-Trait Anxiety Inventory (STAI-S) | At baseline (admission for labor) and immediately after the intervention
  Maternal anxiety will be measured using the State subscale of the State-Trait Anxiety Inventory (STAI-S).
  Scores range from 20 to 80, with higher scores indicating greater anxiety. Mean scores will be analysed at each assessment point.
Childbirth satisfaction as measured by the Childbirth Experience Questionnaire (CEQ) | Within 48 hours postpartum
  Childbirth satisfaction will be assessed using the Childbirth Experience Questionnaire (CEQ).
  Total and domain scores will be calculated according to the scoring guidelines, with higher scores indicating greater satisfaction.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Birckhead B, Khalil C, Liu X, Conovitz S, Rizzo A, Danovitch I, Bullock K, Spiegel B. Recommendations for Methodology of Virtual Reality Clinical Trials in Health Care by an International Working Group: Iterative Study. JMIR Ment Health. 2019 Jan 31;6(1):e11973. doi: 10.2196/11973. PMID 30702436